CLINICAL TRIAL: NCT02426619
Title: A Randomized Clinical Trial on the Use of Sodium Fluoride Varnish and Silver Diamine Fluoride Solution for Arresting Active Dental Caries in Preschool Children
Brief Title: Arresting Active Dental Caries in Preschool Children by Topical Fluorides
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW12-490
Record Dates: First submitted 2014-11-17; First posted 2015-04-27 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SDF regular (Experimental): 3 applications of a 30% SDF solution will be applied onto the surface of dental caries lesions by a small brush regularly once a year
  Interventions: Device: SDF solution
- SDF intensive (Experimental): 3 applications of a 30% SDF solution will be applied onto the surface of dental caries lesions by a small brush at weekly interval at baseline
  Interventions: Device: SDF solution
- NaF varnish (Active Comparator): 3 applications of a 5% NaF varnish will be applied onto the surface of dental caries lesions by a small brush at weekly interval at baseline
  Interventions: Device: NaF varnish

INTERVENTIONS:
Device: SDF solution — around 1 mL of 30% silver diammine fluoride (SDF) solution is placed in a small disposable container and a small brush will be used to apply a very small quantity of the solution onto the surface of the dental caries lesion in the tooth
  Other Names: silver diammine fluoride solution
  Arms: SDF intensive; SDF regular
Device: NaF varnish — around 1 mL of 5% NaF (sodium fluoride) varnish is placed in a small disposable container and a small brush will be used to apply a very small quantity of the solution onto the surface of the dental caries lesion in the tooth
  Other Names: sodium fluoride varnish
  Arms: NaF varnish

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of three topical fluoride application protocols, namely three applications of a 30% SDF solution at yearly or weekly interval and three applications of a 5% NaF varnish at weekly interval, in arresting dental caries in the primary teeth of preschool children over 30 months.

DETAILED DESCRIPTION:
This randomized clinical trial aims to compare the effectiveness of three topical fluoride application protocols, namely three applications of a 30% SDF solution at yearly or weekly interval and three applications of a 5% NaF varnish at weekly interval, in arresting dental caries in the primary teeth of preschool children over 30 months.

Preschool children attending the first year of the kindergartens will be invited to join this study. An invitation letter will be sent to the parents explaining the purpose and procedures of this study. Parental consent will be sought. Generally healthy children who have at least one tooth with untreated caries into dentine will be invited to participate and they will be followed for 30 months.

Dental clinical examination of the children will be conducted by a calibrated dentist in the kindergarten. Tooth and oral hygiene condition will be recorded. A parental questionnaire will be administered at baseline and at the 30-month follow-up visits regarding their children's socio-economic background and oral health related behaviours. The questionnaire will also assess parental satisfaction with their child's oral health and dental aesthetics.

All active dental caries lesions of the participant children will be treated if possible. The children will be categorized as having a high or a low caries rate. They will then be allocated by a stratified randomization method to one of the three study groups:

Group A - 3 applications of a 30% SDF solution at yearly interval Group B - 3 applications of a 30% SDF solution at weekly interval Group C - 3 applications of a 5% NaF varnish at weekly interval

A dental operator who is not involved in the examination of the child will apply the fluoride agents. Follow-up oral examinations will be conducted every 6 months in the kindergartens for 30 months. The status of the treated teeth and any possible side/adverse effects will be recorded in the follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy children who have at least one tooth with untreated caries into dentine

Exclusion Criteria:

* Children who have major systemic diseases or on long-term medication, are uncooperative or refuse the treatment will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
change in hardness of dental caries lesion | baseline and 30 months
  change from a soft active dental caries lesion at baseline to a hardened arrested caries lesion upon gentle probing with a dental explorer at the evaluation is regarded as a positive treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Edward CM Lo, BDS, PhD, Principal Investigator — Faculty of Dentistry, University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China